CLINICAL TRIAL: NCT02284698
Title: Corneal Ulcer Prevention Through Health Education
Acronym: CUP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aravind Eye Care System (Other)
Collaborators: Proctor Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. M.Srinivasan, Prinicpal Investigator, Aravind Eye Care System
Other Study IDs: Aravind-RES2013064CLI
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study Group: Study Group will have the field workers and active health education with referral mechanism
  Interventions: Other: Health Education
- Control Group: Control group will not have field workers and active health education. They will follow routine health care
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Health Education — Heath education will be given through awareness creation & pamphlet distribution

SUMMARY:
A community-randomized trial comparing villages randomized to receive an intervention consisting of a trained community health volunteer who brings patients to the nearest Vision Centers or Primary Health Care Centers for treatment after diagnosing a corneal abrasion to control villages receiving no additional intervention. The primary outcome of corneal ulcer will be measured by baseline and annual population-based census performed in both intervention and control villages by masked examiners from baseline to 24 months. Each resident in the village will be asked about their ocular history and, if suspected of having a corneal ulcer, will be examined for evidence of a corneal opacity. Annual visits will occur, coinciding with the end of the harvest season. In villages randomized to intervention, an active promotion campaign will be undertaken to urge residents to notify the village eye health worker within 24 hours of ocular trauma. In control villages, abrasions and ulcers will be treated if they present to a clinic or are found during the annual monitoring visits, but active promotion of corneal abrasion care will not be offered.

DETAILED DESCRIPTION:
Research Question: Can the investigators prevent corneal ulcers on a mass scale?

Aim 1: To determine whether diagnosis and prophylaxis of corneal abrasions by village health workers will reduce the incidence of corneal ulceration in rural South India. The investigators hypothesize that communities in which village eye health workers are available to diagnose and prophylax corneal abrasions will have a significantly lower incidence of corneal ulceration compared to communities without this service.

Aim 2: To determine the cost-effectiveness of a village eye worker program to prevent corneal ulcers. The investigators hypothesize that preventing corneal ulcers through a village eye worker program will be more cost-effective than the current standard of treating corneal ulcers after patients present at health care facilities.

Aim 3: To determine the incidence of corneal ulceration in this South Indian population. The investigators anticipate that the incidence of ulcers is lower than estimated in our 1995 incidence survey, but still far higher than that observed in the developed world.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a corneal abrasion
* Willingness to be treated with topical antibiotic and antifungal ointments 3 times a day for 3 days
* Appropriate consent

Exclusion Criteria:

* Evidence of a corneal ulcer
* Evidence of other acute eye disease requiring urgent care
* Known allergy to study medications
* Not willing to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 42 villages eligible for the study will comprise a total population of 98,207
Sampling Method: Probability Sample
Enrollment: 98207 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Corneal Ulcer | 2 years
  The primary outcome for the trial will be the incidence of corneal ulceration in the two study arms as measured by field examination.

REFERENCES:
- [Derived] Srinivasan M, Ravilla T, Vijayakumar V, Yesunesan D, Mani I, Whitcher JP, Oldenburg CE, O'Brien KS, Lietman TM, Keenan JD. Community Health Workers for Prevention of Corneal Ulcers in South India: A Cluster-Randomized Trial. Am J Ophthalmol. 2022 May;237:259-266. doi: 10.1016/j.ajo.2021.12.010. Epub 2021 Dec 21. PMID 34942106